CLINICAL TRIAL: NCT04723017
Title: Development and Validation of Perioperative Hypoxemia Using Clinical Big Data and Deep Learning Technique in Pediatric Patients
Brief Title: Perioperative Hypoxemia in Pediatrics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, professor, Seoul National University Hospital
Other Study IDs: 2011-208-1179
Record Dates: First submitted 2021-01-21; First posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Hypoxemia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Retrospective analysis cohort — We analyze pre-existing data base and develop machine-learning-based system that predicts the risk of hypoxemia
Other: Prospective validation cohort — We validate our model to predict the risk of hypoxemia to prospective cohort

SUMMARY:
The primary aim was to develop and validation of perioperative hypoxemia using clinical big data and deep learning technique in pediatric patients

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients undergoing general or spinal anesthesia and monitored anesthesia care

Exclusion Criteria:

* none

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric patients
Sampling Method: Non-Probability Sample
Enrollment: 17000 (Estimated)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
hypoxemia | from induction of anesthesia to end of operation, about 3 hours
  pulse oximetry desaturation below 95%

CONTACTS AND LOCATIONS:
Locations (1):
- Hee-Soo Kim, Seoul, Soul-t'ukpyolsi, South Korea